CLINICAL TRIAL: NCT02522598
Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate the Analgesic Efficacy and Safety of VVZ-149 Injection for Post-operative Pain Following Laparoscopic-assisted Gastrectomy in Early Gastric Cancer Patients
Brief Title: Evaluate the Analgesic Efficacy and Safety of VVZ-149 Injection for Post-operative Pain Following Gastrectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vivozon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT-VVZ149-04
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VVZ-149 injection (Experimental): VVZ-149 Injections will be mixed with saline,then intravenous infusion for 8hr. The drug product will be administered with a loading dose of 1.8 mg/kg for 0.5 hour followed by a maintenance dose of 1.3 mg/kg/h for 7.5 hours.
  Interventions: Drug: VVZ-149 injections
- Placebo (Placebo Comparator): placebo group will receive an water for injection the same volume and period of experimental group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VVZ-149 injections — Colorless, transparent liquid in water for injection
  Other Names: VVZ-149 injection or water for injection
  Arms: VVZ-149 injection
Drug: Placebo — water for injection
  Other Names: VVZ-149 injection or water for injection
  Arms: Placebo

SUMMARY:
VVZ-149 is a novel analgesic drug candidate that shows a potential analgesic activity inhibiting GlyT2 and 5HT2A simultaneously. These target receptors have been known to play important roles in induction and transmission of pain signals. There have been many efforts to develop selective drugs to treat pain, but usually unsuccessful due to the lack of efficacy or limitations of single-target approach for new drug discovery. VVZ-149 is expected to be a dual-target drug, demonstrated having a potential synergism between GlyT2 and 5HT2A to maximize an antinociceptive effect in the in vivo animal models. In Phase 1 conducted among healthy subjects, safety and tolerability were confirmed. Phase 2 was designed as a randomized, double-blind, parallel-group, placebo-controlled trial to evaluate the efficacy and safety of the analgesic drug VVZ-149 injection.

DETAILED DESCRIPTION:
VVZ-149 is a dual antagonist of GlyT2 and 5HT2A. GlyT2 blockage increases inhibitory synaptic transmission by glycine in the spinal cord, resulting in a reduction of pain transmissions to the brain. 5HT2A blockage decreases descending serotonergic facilitatory modulation on pain transmission by the brain and reduces nociceptor activation in peripheral nerves, which are primary sources of pain in post-surgical pain. VVZ-149 has been shown to have comparable efficacy to morphine in well controlled (blind, complete randomization with a positive control) animal studies using rat models of post-operative pain and formalin-induced pain. The PK/PD study in animals indicates that therapeutic plasma concentration in human subjects will be 600-1,900 ng/ml. A clinical Phase 1 study performed in healthy subjects has shown no clinically significant adverse events up to a plasma concentration level of 3,261 ng/ml other than brief symptoms of mild nausea or dizziness, and mild somnolence when the plasma exposure level is more than 2,000 ng/ml.

ELIGIBILITY:
Inclusion Criteria:

1. Patient between the ages of 25 and 70 years old
2. Male patient, in the case of female patient, postmenopausal women, or women physically incapable of childbearing
3. Minimal pain intensity (NRS) of ≥5 at initial post-operative measurement.
4. Subject who underwent surgery specially for the clinical study
5. Ability to provide written informed consent prior to any study procedures.
6. Ability to understand study procedures and communicate clearly with the investigator and staff.
7. Subjects with body weight under 100kg and body mass index (BMI) level lower than 35 kg/m2, inclusive

Exclusion Criteria:

< Surgical Factors >

1. Emergency or unplanned surgery.
2. Repeat operation (e.g., previous surgery within 30 days for same condition).
3. Cancer-related condition causing preoperative pain in site of surgery.

   < Subject Characteristics >
4. Women with childbearing potential, Women who are pregnant or breastfeeding.
5. Chronic pain diagnosis (e.g., ongoing pain at baseline with NRS ≥ 4/10).
6. Unstable or poorly controlled psychiatric condition (e.g., untreated PTSD, anxiety, or depression). Subjects who take stable doses (same dose >30 days) of antidepressants and anti-anxiety drugs may be included.
7. Unstable or acute medical condition (e.g., unstable angina, congestive heart failure, renal failure, hepatic failure, AIDS).
8. Subjects who have long PR (>200msec) or prolonged QTc (> 450msec) at Screening

   < Drug, Alcohol, and Pharmacological Considerations >
9. History of alcohol, opiate or other drug abuse or dependence within 12 months prior to Screening .
10. Ongoing or recent (within 30 days prior to surgery) use of steroids, opioids, or antipsychotics.
11. Alcohol consumption within 24 hours of surgery.
12. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) or acetaminophen within 24 hours of surgery.
13. Use of herbal agents or nutraceuticals (i.e., chaparral, comfrey, germander, jin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian) within 7 days prior to surgery.

    < Anesthetic and Other Exclusion Considerations >
14. Use of neuraxial or regional anesthesia related to the surgery.
15. Use of ketamine, gabapentin, pregabalin, or lidocaine (>1 mg/kg) intra or peri-operatively, or within 24 hours of surgery.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change of Numerical Rating Scale using(NRS) a 10-point scale upto 24hr | prior to administration, at 15 min, 30 min, 1, 2, 4, 6, 8, 10, 24 hours post-dose

SECONDARY OUTCOMES:
Difference of Opioid Consumption between Study Groups | 0-2, 2-4, 4-6, 6-8, 8-12, 12-16, 16-24 hours post-dose
Change of Pain Relief (PR) using a 6-point categorical scale upto 24hours | 15min, 30 min, 1, 2, 4, 6, 8, 10, 20, 24 hours post-dose
Pain Intensity Difference (PID) upto 24hours | pre-administration of investigational drug and at 15 min, 30 min, 1, 2, 4, 6, 8, 10, 24 hr post dosing
  Pain Intensity using a 10-point categorical scale
Sum Pain Intensity Difference over 8hr post- dose (SPID-8) | pre-administration of investigational drug and at 15 min, 30 min, 1, 2, 4, 6, 8, 10, 24 hr post dosing
global measurement of patient satisfaction | 8, 24 hours after dosing
Change of Incidence of Postoperative Nausea and Vomiting(PONV) upto 24hr | pre-administration of investigational drug and at 15 min, 30 min, 1, 2, 4, 6, 8, 10, 24 hours post dosing
Change of Richmond Agitation-Sedation Scale(RASS) upto 24hr | pre-administration of investigational drug and at 15 min, 30 min, 1, 2, 4, 6, 8, 10, 24 hours post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Seonjun Bae, MD, PhD, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea